CLINICAL TRIAL: NCT02005536
Title: Immunogenicity and Safety of IMOVAX POLIO® Subcutaneous as a Booster Given in Pre-school Age Children in Japan
Brief Title: Study of IMOVAX POLIO® Subcutaneous as a Booster Vaccine in Pre-school Age Children in Japan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPV46 (EFC13614); U1111-1143-8561 (Other: WHO)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Poliomyelitis; Polio
Keywords: Poliomyelitis; Poliovirus; Polio; IMOVAX POLIO®; Inactivated polio vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants will receive one booster dose of SP059 (IMOVAX POLIO®)
  Interventions: Biological: IMOVAX POLIO®: Inactive Poliovirus Vaccine

INTERVENTIONS:
Biological: IMOVAX POLIO®: Inactive Poliovirus Vaccine — 0.5 mL, Subcutaneous
  Other Names: SP059; IMOVAX POLIO®

SUMMARY:
The aim of the study is to assess the immunogenicity of SP059 (IMOVAX POLIO®: Inactive Poliovirus Vaccine) vaccine against poliovirus and safety after fifth dose.

Primary Objective:

* To investigate the booster vaccine response rate against poliovirus types 1, 2 and 3 one month following the vaccination dose with SP059 as 2nd booster

Secondary Objectives:

* To investigate seroprotection rates (percentage of subjects presenting poliovirus neutralizing antibody titers above 1:8 (1/dil.) at pre- and post-booster time points, Geometric mean titers (GMT) at pre- and post-booster time points and geometric mean of individual titer ratio (GMTR).
* To investigate the safety after dosing of SP059 as 2nd booster.

DETAILED DESCRIPTION:
Participants will receive one dose of SP059 (at Visit 1) as a booster vaccination at an age from 4 to 6 years. They will be assessed for immunogenicity at baseline (pre-vaccination) and at 4-6 weeks post- vaccination.

Safety data including serious adverse events (SAEs) after vaccination will be collected during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 to 6 years inclusive on the day of inclusion
* Subjects who received 4 times an IPV-containing vaccine (DTaP-IPV or IPV) during first (3 doses) and second year of life (one dose)
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Fever ≥ 37.5°C (axillary temperature) on the day of inclusion
* Any serious disease whether acute or chronic
* Past or current medical history of Guillain-Barre syndrome, acute thrombocytopenic purpura or encephalopathy
* History of poliomyelitis infection
* History of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* History of anaphylaxis or allergy to any of the study vaccine components
* Congenital or current/previous acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Participation in another clinical trial within 6 months before the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Received oral or injected antibiotic therapy within the 72 hours prior to any blood draw
* Received antipyretics/analgesics/Non-steroidal anti-inflammatory drugs (considered as a single category) within 4 hours prior to vaccination
* Blood or blood-derived products received in the past or current or planned administration during the trial (including immunoglobulins)
* Any vaccination with live vaccines within the past 27 days preceding the trial vaccination
* Any vaccination with inactivated vaccines within the past 6 days preceding the trial vaccination
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or HIV infection
* Subject ineligible according to the Investigator's clinical judgment.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi
Locations (4):
- Japan (4):
  - Fukuoka
  - Hokkaido
  - Mie
  - Tokyo

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 02 December 2013 to 28 April 2014 at 4 Clinical trial centers in Japan.
Pre-assignment Details: A total of 60 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated. A subject with an exclusion criteria was later discovered and was excluded in the per-protocol analysis set.
Groups:
- IMOVAX POLIO® Vaccine Group: Participants received a single booster dose of IMOVAX POLIO® vaccine on Day 0.
Period: Overall Study
Arm/Group | IMOVAX POLIO® Vaccine Group
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 35
Region of Enrollment [Number; unit: Participants]
  Japan | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Booster Responses Against Polio Antigens Following Vaccination With IMOVAX POLIO®
Description: A booster response was defined as a 4-fold increase from pre-booster to post-booster vaccination. Anti-polio virus antibodies were assessed by virus neutralization assay.
Time Frame: Day 28 post-vaccination
Population: Anti-polio booster response was assessed in the per-protocol analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 59
Percentage of participants
  Anti-polio 1 | 78.0
  Anti-polio 2 | 78.0
  Anti-polio 3 | 79.7

2. Secondary Outcome: Geometric Mean Titers of Vaccine Antigens Before and After Vaccination With IMOVAX POLIO®
Description: Anti-polio virus antibodies were assessed by virus neutralization assay.
Time Frame: Day 0 (pre-booster vaccination) and Day 28 post-booster vaccination
Population: Geometric mean titers was assessed in the per-protocol analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 59
Titers
  Anti-polio 1 (pre-vaccination) | 312.6 [241.8 to 404.1]
  Anti-polio 1 (post-vaccination) | 3794.9 [3011.5 to 4782.1]
  Anti-polio 2 (pre-vaccination) | 795.4 [591.8 to 1069.1]
  Ant-polio 2 (post-vaccination) | 9213.2 [6754.5 to 12567.0]
  Anti-polio 3 (pre-vaccination) | 314.5 [219.5 to 450.4]
  Anti-polio 3 (post-vaccination) | 5242.1 [3912.9 to 7022.9]

3. Secondary Outcome: Percentage of Participants With Seroprotection Against Polio Antigens Before and After Booster Vaccination With IMOVAX POLIO®
Description: Seroprotection was defined as a titer of ≥ 8 (1/dil) pre-booster or post-booster vaccination. Anti-polio virus antibodies were assessed by virus neutralization assay
Time Frame: Day 0 (pre-booster vaccination) and Day 28 post-booster vaccination
Population: Anti-polio booster response was assessed in the per-protocol analysis set.
Measure: Number; unit: Percentage of participants
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 59
Percentage of participants
  Anti-polio 1 (pre-vaccination) | 100
  Anti-polio 1 (post-vaccination) | 100
  Anti -polio 2 (pre-vaccination) | 100
  Anti-polio 2 (post-vaccination) | 100
  Anti-polio 3 (pre-vaccination) | 98.3
  Anti-polio 3 (post-vaccination) | 100

4. Secondary Outcome: Geometric Mean of Individual Titer Ratios of Vaccine Antigens Following Booster Vaccination With IMOVAX POLIO®
Description: Anti-polio virus anti-bodies were assessed by virus neutralization assay. The geometric mean titer ratio is the post-booster to pre-booster geometric mean ratio values.
Time Frame: Day 28 post-booster vaccination
Population: Geometric mean of individual titer ratios were assessed in the per-protocol analysis set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer Ratio
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 59
Titer Ratio
  Anti-polio 1 | 12.1 [8.5 to 17.4]
  Anti-polio 2 | 11.6 [7.7 to 17.5]
  Anti-polio 3 | 16.7 [9.8 to 28.4]

5. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reaction Following Booster Vaccination With IMOVAX POLIO®
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Fever, Headache, Malaise, Myalgia. Grade 3 was defined as incapacitating, unable to perform usual activities for Pain; diameter ≥ 50 mm for Erythema and Swelling; Temperature ≥ 39.0°C for Fever; and significant, prevents daily activity for Headache, Malaise, and Myalgia.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all participants who received study vaccine (Safety Analysis Set).
Measure: Number; unit: Number of participants
Arm/Group | IMOVAX POLIO® Vaccine Group
Number analyzed (Participants) | 60
Number of participants
  Any Injection-site Pain | 13
  Grade 3 Injection-site Pain | 0
  Any Injection-site Erythema | 41
  Grade 3 Injection-site Erythema | 1
  Any Injection-site Swelling | 21
  Grade 3 Injection-site Swelling | 0
  Any Fever | 8
  Grade 3 Fever | 2
  Any Headache | 4
  Grade 3 Headache | 0
  Any Malaise | 18
  Grade 3 Malaise | 0
  Any Myalgia | 1
  Grade 3 Myalgia | 0

ADVERSE EVENTS:
Time Frame: Safety was evaluated from Day 0 (post-booster vaccination) up to Day 28 post-booster vaccination.
Description: The total number (47) reporting other adverse events at the 5% frequency are those participants with solicited injection site and systemic reactions.
Arm/Group | IMOVAX POLIO® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 47/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMOVAX POLIO® Vaccine Group (N=60)
Injection Site Erythema (General disorders) | 41
Injection Site Pain (General disorders) | 13
Injection Site Swelling (General disorders) | 21
Malaise (General disorders) | 18
Headache (Nervous system disorders) | 4
Fever (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 4
Gastroenterities (Infections and infestations) | 3
Varicella (Infections and infestations) | 3
Diarrhoea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications